CLINICAL TRIAL: NCT03272568
Title: A Feasibility Trial Using Extended Half Life Factor Products in the Reduction of Menstrual Bleeding in Symptomatic Hemophilia A and B Carriers
Brief Title: Extended Half Life Factor (EHF) Products For Heavy Menstrual Bleeding in Hemophilia Carriers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bioverativ Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Robert Sidonio, Assistant Professor of Pediatrics, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00095067
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia; Menstrual Flow Excessive
Keywords: Extended Life Plasma Derived Factor Products; Female hemophilia A and B carriers; Menorrhagia
MeSH Terms: conditions — Hemophilia A; Menorrhagia | interventions — factor VIII-Fc fusion protein; factor IX Fc fusion protein

STUDY DESIGN:
Intervention Model Description: During interventional portion of the study, participants will be infused with either Eloctate (hemophilia A carriers) or Alprolix (hemophilia B carriers) to maintain FVIII or FIX >48hours. Five out of the 16 enrolled patients will self-perform a hemoglobin check every other day using a novel device Anemocheck during 2 consecutive menstrual cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Hemophilia A symptomatic female carriers (Experimental): Hemophilia A symptomatic female carriers with a baseline FVIII activity of ≤60% receive recombinant FVIII Fc fusion product Eloctate.
  Some of participants will be taught to perform a hemoglobin check using a patient-operated diagnostic device for anemia AnemoCheck every other day during 2 consecutive menstrual cycles.
  Interventions: Drug: Recombinant FVIII Fc fusion product Eloctate; Device: Patient-operated diagnostic device for anemia AnemoCheck.
- Hemophilia B symptomatic female carriers (Experimental): Hemophilia B symptomatic female carriers with a baseline FIX activity of ≤60% receive recombinant FIX Fc fusion product Alprolix.
  Some of participants will be taught to perform a hemoglobin check using a patient-operated diagnostic device for anemia AnemoCheck every other day during 2 consecutive menstrual cycles.
  Interventions: Drug: Recombinant FIX Fc fusion product Alprolix; Device: Patient-operated diagnostic device for anemia AnemoCheck.

INTERVENTIONS:
Drug: Recombinant FVIII Fc fusion product Eloctate — Subjects will get FVIII activity corrected from the baseline level to 100-150% with Eloctate on the first day of menstruation at the beginning of the study interventional phase. The first dose of the drug will be given in the clinics via slow injection into a vein (infusion). A short assessment of pharmacokinetics (PK) (4 time-points blood draw: 15 min, 2 hours, 4 hours, 20 hours after the infusion) will be performed to assist with subsequent dosing. 2 total doses of Eloctate likely to be given on day 1 and 3 of menstrual period. The subject will then receive three additional PK-adjusted monthly doses of Eloctate (with no less than 21 days interval).
  Other Names: Eloctate
  Arms: Hemophilia A symptomatic female carriers
Drug: Recombinant FIX Fc fusion product Alprolix — Subjects will get FIX activity corrected from the baseline level to 100-150% with Alprolix on the first day of menstruation at the beginning of the study interventional phase. The first dose of the drug will be given in the clinics via slow injection into a vein (infusion). A short assessment of pharmacokinetics (PK) (4 time-points blood draw: 15 min, 4 hours, 48 hours, 72 hours after the infusion) will be performed (by home nursing or local lab) to assist with subsequent dosing. Single dose of Alprolix likely to be given on day 1 of menstrual period. The subject will then receive three additional PK-adjusted monthly doses of Alprolix (with no less than 21 days interval).
  Other Names: Alprolix
  Arms: Hemophilia B symptomatic female carriers
Device: Patient-operated diagnostic device for anemia AnemoCheck. — Each AnemoCheck test kit enables patients to check hemoglobin levels by pricking their finger to draw 5 μL of blood into a capillary tube, inserting that tube into a larger tube with a pre-filled chemical solution, mixing, waiting one minute, and assessing the color change of the solution using a reference color scale card included with the kit. The test is able to subjectively differentiate low, medium and high levels of hemoglobin to diagnose anemia at home. Study participants are taught to perform a hemoglobin check every other day using Anemocheck during 2 consecutive menstrual cycles. In addition they will have hemoglobin level obtained locally (LabCorp) drawn within 4-6 hours for comparison and correlation.
  Other Names: AnemoCheck

SUMMARY:
The purpose of this feasibility study is to find out if two clotting factor products, Eloctate [hemophilia A] and Alprolix [hemophilia B], can reduce the amount of menstrual bleeding in female hemophilia A and B carriers (14 years of age or older) who have severe or heavy bleeding. These products are FDA-approved for use in males with hemophilia A and B to prevent and treat bleeding. They are not approved specifically to reduce menstrual bleeding, but may be useful for this purpose. Both products have an "extended half life" which means they circulate in the body longer than other FVIII or FIX products. The study team will gather additional information about the safety of these drugs and how well they work. The results of this feasibility study will provide information for an upcoming larger study.

DETAILED DESCRIPTION:
Hemophilia A or B is caused by defects in the factor VIII or IX gene, respectively, of which is located on the X chromosome. This disorder exhibits X-linked inheritance, in which primarily males, with a single X chromosome, are affected and females, with two X chromosomes, are heterozygotes, or carriers. Hemophilia carriers show a wide distribution of factor VIII or IX levels with a mean of 50%, which overlaps the distribution of non-carrier women.

Heavy menstrual bleeding is defined as menstrual bleeding that lasts more than 7 days or more specifically as the loss of more than 80cc of blood per cycle. Management is critical as it can lead to iron deficiency anemia, lead to school absence and affects the general quality of life. There are multiple options to control or reduce menstrual bleeding in hemophilia A and B carriers, they include but not limited to the following options: Antifibrinolytics (Aminocaproic acid, Tranexamic acid), Synthetic desmopressin (DDAVP, SQ or IN) or hormonal therapies (Combined oral contraceptives, Progestin only options, IUD, etc).

The use of recombinant factor replacement has been poorly studied and limited by a relatively short half-life in relation to the typical length of a menstrual period. The purpose of this feasibility study is to find out if two clotting factor products, Eloctate [hemophilia A] and Alprolix [hemophilia B], can reduce the amount of menstrual bleeding in female hemophilia A and B carriers (14 years of age or older) who have severe or heavy bleeding. These products are FDA-approved for use in males with hemophilia A and B to prevent and treat bleeding. They are not approved specifically to reduce menstrual bleeding, but may be useful for this purpose. Both products have an "extended half life" which means they circulate in the body longer than other FVIII or FIX products. The study team will gather additional information about the safety of these drugs and how well they work. Five out of the 16 anticipated enrolled patients will be approach to request participation in the exploratory aim in which the subject is taught to perform a hemoglobin check (CBC) every other day using a novel point of care device (Anemocheck) during 2 consecutive menstrual cycles. In addition, they will have CBCs drawn within 4-6 hours for comparison and correlation. The study team will also correlate symptoms of heavy menstrual bleeding with a 2grams drop in the hemoglobin. All the results of this study will provide information for an upcoming larger study.

ELIGIBILITY:
Inclusion Criteria:

* Females of reproductive age who experience monthly menstrual bleedings
* Female Hemophilia A or B carrier (heterozygote, lyonized or Turner's Syndrome)
* FVIII or FIX activity ≤60% at time of the study
* Baseline Pictorial Bleeding Assessment Chart >150 mean at time of recruitment
* Negative pregnancy test at time of enrollment
* Both female and her male partner have agreed to use an acceptable barrier method of birth control (e.g., diaphragm, cervical cap, male condom, female condom, and spermicidal foam, sponges, and film) throughout the duration of this study (for sexually active participants)

Exclusion Criteria:

* Has not reached menarche
* Menopause: natural or induced by surgical/medical treatment
* Pregnant or breasfeeding
* Female or her male partner refuses to use barrier method of birth control (for sexually active)
* Current use of any of the following contraceptives (copper IUD, oral combined, Progestin-only including but not limited to: Provera, Aygestin, Nexplanon, Implanon, Depo Provera, Mirena IUD)
* VWF:Ag or VWF:RCo <40%
* Diagnosis of a qualitative platelet disorder
* Personal history of thrombosis or superficial thrombosis
* First degree relative with a history of thrombosis
* Personal history of concomitant bleeding or clotting disorder
* Cigarette smoker
* Willing to avoid taking an anti-fibrinolytic agent (amicar, transexamic acid, lysteda) during the trial

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 3 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in menstrual bleeding measured by the Pictorial Bleeding Assessment Chart (PBAC). | Monthly throughout study duration for 7 months
  Menstrual loss is tracked via paper and electronic PBAC, calculated via visual interpretation centrally and correlated to the ability of a participant to correctly assign pad or tampon saturation. The PBAC will be estimated (mean) over the three-month intervention period to assess if 30% reduction in menstrual bleeding was achieved. PBAC is a semi-quantitative, self-administered pictorial tool. The total score is calculated by adding up the sum of all scores for the tampons or pads used, with a score greater than 150 having an 86% sensitivity and 89% specificity for heavy menstrual bleeding (HMB). Possible range is dependent on quantitative and qualitative amount of bleeding during menstruation:
  * For tampons: 0.5-1 for lightly stained, 1-4 for moderately soiled and 4-12 for completely saturated tampons.
  * For pads: 1 for lightly stained, 2-6 for moderately soiled and 4-15 for completely saturated pads.
  * Clots were given a score of 1 for small and 5 for large clots.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS-43) score. | Monthly, prior to the beginning of each menstrual cycle either by phone or in person for the study duration of 7 months.
  To determine whether the use of the study drugs leads to a significant improvement in Quality of Life (QOL) the study establishes a baseline QOL and measures change monthly and 6-month change. The PROMIS 43 profile is a QOL assessment tool of 43 questions from 9 health domains and 10 questions focused on sexual health. The PROMIS assesses patient reported outcomes in three major categories: physical health, mental health, and social health. Each item has five response options except for the Pain Intensity item which has eleven options.A raw score is created from each short form. To find the total raw score the values of the response to each question are summed up within each domain. The applicable score conversion table translates the total raw score into standardized T-score that is reported as the final score.
Change in Short Form 36 (SF-36) score. | Monthly, prior to the beginning of each menstrual cycle either by phone or in person for the study duration of 7 months
  To determine whether the study treatment leads to a clinically significant improvement in Quality of Life (QOL) the study team establishes a baseline quality of life and measures change monthly as well as 6-month change in SF-36. SF-36 is a a 36-item patient reported survey of health consisting of 8 scaled scores with a lower score indicating disability in the one of the 8 sections or domains.The scoring system for the SF-36 is relatively complex and generates subscale scores for physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role-limitations due to emotional problems, and mental health. Two summary scores can also be derived from the SF-36: the physical component summary and the mental component summary.
Change in Menorrhagia Impact Questionnaire (MIQ) score. | Monthly, prior to the beginning of each menstrual cycle either by phone or in person for the study duration of 7 months
  The MIQ consists of six individual measures or items. The first 4 items are evaluated by using 4-point (item 1) or 5-point (items 2-4) response scales. No summative scale is derived for item 5 as it serves as a descriptive tool to characterize limitations of specific activities and is viewed as supporting information for items 2-4. Item 6 represents a global assessment (impact, degree, and meaningfulness) of the change in menstrual bleeding lost (MBL) when compared to the previous period. Impact response options included a 0 ('almost the same'), 1 ('better'), or 2 ('worse'). If a change is reported, then a 7-point rating scale is used to specify the degree of improvement (item 6a) or worsening (item 6b). Finally, item 6c (meaningfulness of change in MBL) provides an overall assessment of the subjective perception of the change in MBL and may be considered an important component of the MIQ.
Number of hypersensitivity reactions. | Througout the interventional phase of the study (visit 4-7 of the study or months 4-7)
  Since Eloctate and Alprolix are biological products, hypersensitivity reactions, including anaphylaxis and anaphylactic reactions, may occur. Nurses and patients will be trained to recognize the signs and symptoms associated with potential hypersensitivity, anaphylactic, and anaphylactoid reactions, and instructed to provide/seek immediate care. Patients/caregivers will receive two alert cards with this information and instructions. For patients with a previous history of a clinically significant hypersensitivity reaction, the site will call the patient 24 hours after each dose to assess the status of the patient. Additional precautions following each of these doses may also be considered including having an extended observation period or IV access prior to dosing.
Accuracy of hemoglobin levels detection by Anemocheck. | Every other day during 2 consecutive menstrual cycles during non-interventional study phase (up to Day 60 of the study).
  Exploratory arm participants will self-perform hemoglobin check using Anemocheck every other day during 2 consecutive menstrual cycles. To determine the feasibility and utility of Anemocheck in the monitoring of hemoglobin during a menstruation, the study team will assess correlation of symptoms of heavy menstrual bleeding with a 2g drop in the hemoglobin detected by Anemocheck, and correlation of hemoglobin level obtained by local Lab (within 4-6 hours).
Change in FVIII level after the first dose of Eloctate. | First visit of interventional study phase (visit 4, day 90 of the study) : 15-30 min, 2 hours, 4 hours, 18-24 hour after infusion.
  An assessment of FVIII level via blood draw will be performed after the first dose of the drug at four time points.
Change in FIX level after the first dose of Alpolix. | First visit of interventional study phase (visit 4, day 90 of the study) : 15-30 min,4 hours,48 hours, and 72 hours after infusion.
  An assessment of FIX level via blood draw will be performed after the first dose of the drug at four time points.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sidonio, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Clinical Research Network, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided